CLINICAL TRIAL: NCT06593184
Title: Efficacy of Trans-spinal Magnetic Stimulation on Functional Mobility in Chronic Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, Professor, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: tsMS_Stroke_Gait
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Stroke Sequelae; Gait Disorders, Neurologic; Stroke
Keywords: Spinal cord; Magnetic Stimulation; Trans-spinal magnetic stimulation; Stroke
MeSH Terms: conditions — Gait Disorders, Neurologic; Stroke

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial, double blinded (therapist/evaluator, patient) Initial evaluation, followed by 10 days of treatment, followed by a re-evaluation immediately after and follow-up 30 days after finishing.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active trans-spinal magnetic stimulation (Experimental): Trans-spinal magnetic stimulation activates afferent spinal roots and increases cortical excitability.
  Interventions: Device: Trans-spinal magnetic stimulation
- Sham trans-spinal magnetic stimulation (Sham Comparator): Treadmill training with masking for trans-spinal magnetic stimulation
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: Trans-spinal magnetic stimulation — Trans-spinal magnetic stimulation activates afferent spinal roots and increases cortical excitability.
  Other Names: tsMS, transcutaneous spinal cord magnetic stimulation
  Arms: Active trans-spinal magnetic stimulation
Device: Sham Comparator — Sham trans-spinal magnetic stimulation involves masking, where the sound of stimulation persists even though no magnetic pulses are delivered
  Arms: Sham trans-spinal magnetic stimulation

SUMMARY:
The goal of this clinical trial is to learn if trans-spinal magnetic stimulation works to treat gait disorders in chronic stroke adults. It will also learn about the safety of trans-spinal magnetic stimulation.

The main questions it aims to answer are:

Does trans-spinal magnetic stimulation enhance chronic stroke participants gait and functional mobility? Does the technique cause any side effects?

Researchers will compare trans-spinal magnetic stimulation to a sham (a look-alike stimulation with no real effect) to see if trans-spinal magnetic stimulation works to treat gait disorders and improve functional mobility.

Participants will:

Receive trans-spinal magnetic stimulation with treadmill training or a sham stimulation with treadmill training every day for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of Stroke by digital or physical imaging or medical report
* Gait impairment
* Stroke with at least 6 months after ictus

Exclusion Criteria:

* Metallic implants in spinal cord
* Major orthopedic/rheumatological disorders
* Incapacity of verbal or non-verbal communication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Functional Mobility | Enrollment (Day 0); End of treatment (2 weeks); Follow-up after 30 days post-treatment
  The Timed-Up and Go (TUG) test is used to evaluate an individual´s capacity to stand up, walk, and sit down. During the test, the participants are timed from the moment they begin to stand up until they are seated again.

SECONDARY OUTCOMES:
Independency level | Enrollment (Day 0); End of treatment (2 weeks); Follow-up after 30 days post-treatment
  Self-reported independence is assessed using the Functional Ambulation Categories (FAC). Scores range from 0 (inability to walk even with external help) to 5 (normal ambulation).
Lower limb motor function | Enrollment (Day 0); End of treatment (2 weeks); Follow-up after 30 days post-treatment
  Motor function of the lower limbs is assessed using the Fugl-Meyer Assessment, where scores range from 0 (indicating the worst motor function) to 28 (indicating normal motor function).
Balance | Enrollment (Day 0); End of treatment (2 weeks); Follow-up after 30 days post-treatment
  Capacity to maintain balance during various tasks is assessed using the Mini Balance Evaluation System (MiniBEST-test). Its scores range from 0 to 28 points. Lower scores indicate poor balance, while higher scores reflect better balance.
Perceived change in treatment | End of treatment (2 weeks)
  Evaluation of how the participant describes the perceived change in their condition since the treatment started, using the Patient Global Impression of Change (PGM). This scale assesses the change in activity limitations, symptoms, emotions, and overall quality of life since the beginning of treatment, ranging from no change or worsening to significant improvement that made a considerable difference. A score of one indicates no change, while a score of seven represents a substantial improvement.
Spasticity | Enrollment (Day 0); End of treatment (2 weeks); Follow-up after 30 days post-treatment
  Tonus disorders will be assessed using the Modified Ashworth Scale, which measures spasticity by grading muscle resistance during passive stretching. The scale ranges from 0 to 4, where 0 indicates no increase in muscle tone, and 4 represents a limb that is rigid in flexion or extension.
Sensory Function | Enrollment (Day 0); End of treatment (2 weeks); Follow-up after 30 days post-treatment
  Assessed using a method inspired by the ASIA scale, evaluating the lower thoracic, mid-thoracic, and lower cervical dermatomes, where a score of 0 indicates absence of sensitivity and 2 indicates normal sensitivity.

CONTACTS AND LOCATIONS:
Locations (3):
- Brazil (3):
  - Federal University of Paraiba, João Pessoa, Paraíba
  - Federal University of Pernambuco, Recife, Pernambuco
  - Federal University of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: Undecided